CLINICAL TRIAL: NCT02430948
Title: Improving Compliance With Medical Testing Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: OGARA CAN-264
Record Dates: First submitted 2014-09-29; First posted 2015-04-30 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Cervical Cancer; Prostate Cancer; Colon Cancer; Lung Cancer
Keywords: Screening; Shared Decision Making
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Support Outreach (Active Comparator): Providers receive standard written screening recommendations and do not receive academic detailing (educational outreach)
  Interventions: Other: Standard support; Other: No academic detailing
- Standard materials and academic detailing (Experimental): Providers receive standard written screening recommendations and receive academic detailing (educational outreach)
  Interventions: Other: Academic detailing; Other: Standard support
- Color-coded materials and no academic detailing (Experimental): Providers receive color-coded written screening recommendations and do not receive academic detailing (educational outreach)
  Interventions: Other: Color-coded materials; Other: No academic detailing
- Color-coded materials and academic detailing (Experimental): Providers receive color-coded written screening recommendations and receive academic detailing (educational outreach)
  Interventions: Other: Color-coded materials; Other: Academic detailing

INTERVENTIONS:
Other: Color-coded materials — A summary of treatment recommendations for each cancer screening is color-coded to indicate the strength and direction of the recommendation
  Arms: Color-coded materials and academic detailing; Color-coded materials and no academic detailing
Other: Academic detailing — Educational outreach to address the rationale and data supporting recommendations for and against screening
  Arms: Color-coded materials and academic detailing; Standard materials and academic detailing
Other: Standard support — Screening recommendations presented in standard format
  Arms: Standard Support Outreach; Standard materials and academic detailing
Other: No academic detailing — Physician receives study orientation for not the academic detailing curriculum
  Arms: Color-coded materials and no academic detailing; Standard Support Outreach

SUMMARY:
The study hypothesis is that clearer visual presentation of guideline recommendations and educational outreach, or academic detailing, can improve guideline compliance. However, it will investigate other aspects of screening-related decision-making, such as provider and patient beliefs about screening, provider-patient communication and patient's willingness to forgo expected testing. The research question is whether educational interventions can decrease non-compliance with screening guidelines for 5 common cancers.

DETAILED DESCRIPTION:
This study is a cluster randomized trial that compares the immediate post-encounter impressions of 12 physicians and 18 of their patients about the discussion of screening for breast, cervical, colorectal, lung and prostate cancer as well as their beliefs about screening efficacy and patient reports of the screening experience. The interventions are educational materials and academic detailing (educational outreach) for providers. The investigators are particularly interested in contrasting the patient and provider recollections, the differential impact on underuse and overuse compliance and whether patient behaviors are consistent with their stated screening plans.

ELIGIBILITY:
Inclusion Criteria:

* Patients: healthy men and women ages 30-89 seeing their primary care provider for routine visit
* Providers: non-pediatric primary care physicians from Mount Sinai Beth Israel or St. Luke's-Roosevelt associated practices

Exclusion Criteria:

* Patient life expectancy of less than 1 year in primary care provider's judgment
* Inability to read and understand English
* Transgender status

Ages: 30 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2014-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Effect of educational intervention on providers' recommendations | Baseline
  Incidence of guidance compliance
Effect of educational intervention on providers' recommendations | 3 months
  Incidence of guidance compliance
Effect of educational intervention on providers' recommendations | 6 months
  Incidence of guidance compliance
Effect of educational intervention on providers' recommendations | 12 months
  Incidence of guidance compliance

SECONDARY OUTCOMES:
Patients' belief in the value of screening | Baseline
  measured by survey to be determined
Patients' belief in the value of screening | 3 months
  measured by survey to be determined
Patients' belief in the value of screening | 6 months
  measured by survey to be determined
Patients' belief in the value of screening | 12 months
  measured by survey to be determined
Patient compliance | Baseline
  measured by self- report in surveys to be determined
Patient compliance | 3 months
  measured by self- report in surveys to be determined
Patient compliance | 6 months
  measured by self- report in surveys to be determined
Patient compliance | 12 months
  measured by self- report in surveys to be determined

CONTACTS AND LOCATIONS:
Overall Officials: James A Talcott, MD SM, Principal Investigator — Mount Sinai Beth Israel
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel, New York, New York
  - St. Luke's-Roosevelt, New York, New York